CLINICAL TRIAL: NCT00419250
Title: A Phase 1, Multi-center, Open-label Study of the Safety and Efficacy of a Stepwise Dose-escalation Schedule of Lenalidomide Monotherapy in Subjects With Relapsed or Refractory B-cell Chronic Lymphocytic Leukemia
Brief Title: A Dose Escalation Study of Lenalidomide in Relapsed or Refractory B-cell Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-CLL-001
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Chronic Lymphocytic Leukemia; Leukemia, B-Cell, Chronic
Keywords: relapsed; refractory; fludarabine; Revlimid; lenalidomide; CLL; B-cell CLL; CC-5013; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Leukemia, B-Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- dose-escalation to 5 mg lenalidomide (len) (Experimental): escalate up to 5 mg once daily / 28-day cycle
  Interventions: Drug: lenalidomide
- dose-escalation to 10 mg lenalidomide (len) (Experimental): escalate up to 10 mg once daily / 28-day cycle
  Interventions: Drug: lenalidomide
- dose-escalation to 15 mg lenalidomide (len) (Experimental): escalate up to 15 mg once daily / 28-day cycle
  Interventions: Drug: lenalidomide
- dose-escalation to 20 mg lenalidomide (len) (Experimental): escalate up to 20 mg once daily / 28-day cycle
  Interventions: Drug: lenalidomide
- dose-escalation to 25 mg lenalidomide (len) (Experimental): escalate up to 25 mg once daily / 28-day cycle
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide
  Other Names: Revlimid, CC-5013
  Arms: dose-escalation to 5 mg lenalidomide (len)
Drug: lenalidomide
  Other Names: Revlimid, CC-5013
  Arms: dose-escalation to 10 mg lenalidomide (len)
Drug: lenalidomide
  Other Names: Revlimid, CC-5013
  Arms: dose-escalation to 15 mg lenalidomide (len)
Drug: lenalidomide
  Other Names: Revlimid, CC-5013
  Arms: dose-escalation to 20 mg lenalidomide (len)
Drug: lenalidomide
  Other Names: Revlimid, CC-5013
  Arms: dose-escalation to 25 mg lenalidomide (len)

SUMMARY:
The purpose of this study is to evaluate the safety of lenalidomide and to define the maximum tolerated escalation dose level (MTEDL) when administered by a stepwise dose-escalation schedule in subjects with relapsed or refractory B-cell CLL.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of B-cell CLL that has relapsed after or is refractory to at least one prior regimen. The prior regimen(s) must have included an alkylating agent and fludarabine (used in combination or separately)
* ECOG < or = 2
* Willing to agree to follow the pregnancy precautions.

Exclusion Criteria:

* Pregnant or nursing women
* Systemic treatment for B-cell CLL within 28 days of study start
* Central nervous system involvement
* History of renal failure requiring dialysis
* Prior treatment with lenalidomide
* Alemtuzumab therapy within 56 days of initiating lenalidomide treatment
* ANC < 1000 / ul
* Platelet count < 50,000 / ul
* Calculated creatinine clearance < 60 mL/min (Cockroft-Gault method)
* AST or ALT > 3.0 x upper limit of normal
* Serum total bilirubin > 2.0 mg/dl
* Neuropathy > or = Grade 2
* Uncontrolled autoimmune hemolytic anemia or thrombocytopenia
* Richter's transformation (active)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-12-01 (Actual); Primary Completion 2010-02-01 (Actual); Study Completion 2010-06-01 (Actual)

PRIMARY OUTCOMES:
Safety | February 2010

SECONDARY OUTCOMES:
Response | February 2010
Duration of response | February 2010
Time to response | February 2010
Progression free survival | February 2010
Overall survival | February 2010
Absolute lymphocyte count | February 2010
Evaluation of minimal residual disease (MRD) by flow cytometry | February 2010

CONTACTS AND LOCATIONS:
Overall Officials: Elayne Lombardy, MD, Study Director — Celgene Corporation; Asher Chanan-Khan, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (35):
- United States (20):
  - Arizona Cancer Center, Tucson, Arizona
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Desert Hematology Oncology Medical Group, Inc., Rancho Mirage, California
  - Baptist Cancer Institute, Jacksonville, Florida
  - Cancer & Blood Disease Center, Lecanto, Florida
  - Northwest Georgia Oncology Centers, PC., Wellstar Health System, Marietta, Georgia
  - Mountain States Tumor Institute, Boise, Idaho
  - Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University Medical center, Indianapolis, Indiana
  - LSU Health Sciences Center, Feist-Weiller Cancer Center, Shreveport, Louisiana
  - Karmanos Cancer Institute/Wayne State University School of Medicine, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Medical College of Cornell University, Division of Hematology & Oncology, New York, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Abington Hematology Oncology Assoc., Inc., Willow Grove, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
- Canada (5):
  - Cross Cancer Institute, Edmonton, Alberta
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Helath Science Centre, London, Ontario
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Germany (4):
  - Uniklinik Köln, Klinik I für Innere Medizin, Klinisches Studienzentrum Hämatologie, Bettenhaus Ebene 04, Raum 001/048, Kerpener Str. 62, Koln
  - Charité, Campus Benjamin Franklin, Medizinische Klinik III, Hindenburgdamm 30, State of Berlin
  - University of Schleswig Holstein, Director Medizinische Klinik II, Campus Kiel, Chemnitzstrasse 33, Kiel
  - University of Ulm, Abteilung Innere Medizin III, Robert-Koch-Strasse 8, Ulm
- Clinica Ematologica- A.O.U. San Martino, Clinica Ematologica Dipartimento di Medicina Interna, Genova, Italy
- Hospital Clinic Provincial de Barcelona, Servicio de Hematología, Institute of Haematology and Oncology, Villaroel, 170, Barcelona, Spain
- Karolinska Universitetssjukhuset, Hematologiskt Centrum, Karolinska Universitetssjukhuset,, Stockholm, Sweden
- United Kingdom (3):
  - St James's Institute of Oncology, Dept. of Haematology, Level 3, Bexley Wing, Beckett Street, Leeds
  - Bart's and the London NHS Trust, St. Bartholomew's Hospital, 7th Floor Gloucester House, Cancer Services, London
  - Christie Hospital NHS Foundation Trust, Haematology and Transplant Unit,, Manchester

REFERENCES:
- [Background] Wendtner CM, Hillmen P, Mahadevan D, Buhler A, Uharek L, Coutre S, Frankfurt O, Bloor A, Bosch F, Furman RR, Kimby E, Gribben JG, Gobbi M, Dreisbach L, Hurd DD, Sekeres MA, Ferrajoli A, Shah S, Zhang J, Moutouh-de Parseval L, Hallek M, Heerema NA, Stilgenbauer S, Chanan-Khan AA. Final results of a multicenter phase 1 study of lenalidomide in patients with relapsed or refractory chronic lymphocytic leukemia. Leuk Lymphoma. 2012 Mar;53(3):417-23. doi: 10.3109/10428194.2011.618232. Epub 2011 Nov 15. PMID 21879809